CLINICAL TRIAL: NCT05850273
Title: Mechanism of Action of Interferon in the Treatment of Myeloproliferative Neoplasms
Acronym: IFN&SMP
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C21-46; 2021-A03067-34 (Other: INSERM)
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Myeloproliferative Neoplasm
Keywords: interferon alpha; Hematopoietic stem cell; mechanism of action
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be sampled and fractionated into different types of progenitors based on CD34, CD38 and CD90 markers, granulocytes, platelets,plasma.
  The progenitor cells will be single cell sequenced or genotyped. Alternatively the progenitor cells will be cultured in vitro. The DNA and RNA will be extracted from granulocytes and platelets respectively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Classical BCR-ABL-negative myeloproliferative neoplasms (MPN) include: Polycythemia Vera (PV), Essential Thrombocythemia (ET) and Primary Myelofibrosis (PMF). They are myeloid malignancies resulting from the transformation of a multipotent hematopoietic stem cell (HSC) caused by mutations activating the JAK2/STAT pathway. The most prevalent mutation is JAK2V617F. Type 1 and Type 2 calreticulin (CALR) and thrombopoietin receptor (MPL) mutations are also observed in ET and PMF. Additional non-MPN mutations affecting different pathways are also found, particularly in PMF, and are involved in disease initiation and/or in phenotypic changes and /or disease progression and/or response to therapy.

There is an obvious and urgent need for an efficient therapy for MPN. In particular, PMF remain without curative treatment, except allogeneic HSC transplantation and JAK inhibitors have limited effects on the disease outcome. Among novel therapeutic approaches, Peg-IFNα2a (IFN) is the most efficient harboring both high rates of hematological responses in JAK2V617F and CALRmut MPN patients and some molecular responses mainly in JAK2V617F patients including deep molecular response (DMR). Nevertheless, several studies, including our own, have demonstrated that the IFN molecular response in CALRmut patients is heterogeneous and overall much lower than in JAK2V617F patients. Moreover, some JAK2V617F MPN patients do not respond to IFN, and DMR is only observed in around 20% of JAK2V617F patients. Finally, long-term treatments are needed (2-5 years) to obtain a DMR, jeopardizing its success due to possible long-term toxicity.

The underlying reasons for failure, drug resistance, heterogeneous molecular response in CALRmut patients and the long delays for DMR in JAK2V617F patients remain unclear, largely because the mechanisms by which IFNα targets MPN malignant clones remain elusive.

Significant improvement of IFN efficacy cannot be achieved without basic and clinical research. Hence our two lines of research are to

* Understand how IFNα specifically targets neoplastic HSCs
* Predicting and improving patient response during IFNα therapy

DETAILED DESCRIPTION:
Classical BCR-ABL-negative myeloproliferative neoplasms (MPN) include: Polycythemia Vera (PV), Essential Thrombocythemia (ET) and Primary Myelofibrosis (PMF). They are myeloid malignancies resulting from the transformation of a multipotent hematopoietic stem cell (HSC) caused by mutations activating the JAK2/STAT pathway. The most prevalent mutation is JAK2V617F. Type 1 and Type 2 calreticulin (CALR) and thrombopoietin receptor (MPL) mutations are also observed in ET and PMF. Additional non-MPN mutations affecting different pathways are also found, particularly in PMF, and are involved in disease initiation and/or in phenotypic changes and /or disease progression and/or response to therapy.

There is an obvious and urgent need for an efficient therapy for MPN. In particular, PMF remain without curative treatment, except allogeneic HSC transplantation and JAK inhibitors have limited effects on the disease outcome. Among novel therapeutic approaches, Peg-IFNα2a (IFN) is the most efficient harboring both high rates of hematological responses in JAK2V617F and CALRmut MPN patients and some molecular responses mainly in JAK2V617F patients including deep molecular response (DMR). Nevertheless, several studies, including our own, have demonstrated that the IFN molecular response in CALRmut patients is heterogeneous and overall much lower than in JAK2V617F patients. Moreover, some JAK2V617F MPN patients do not respond to IFN, and DMR is only observed in around 20% of JAK2V617F patients. Finally, long-term treatments are needed (2-5 years) to obtain a DMR, jeopardizing its success due to possible long-term toxicity.

The underlying reasons for failure, drug resistance, heterogeneous molecular response in CALRmut patients and the long delays for DMR in JAK2V617F patients remain unclear, largely because the mechanisms by which IFNα targets MPN malignant clones remain elusive.

Significant improvement of IFN efficacy cannot be achieved without basic and clinical research. Hence our two lines of research are to

* Understand how IFNα specifically targets neoplastic HSCs
* Predicting and improving patient response during IFNα therapy

The main objective from the basic point of view is to draw the clonal architecture of the mutated cells of the patients during IFN treatment to provide a better understanding of the mechanism of action of IFN in MPN: namely how and at what level of hematopoietic differentiation the IFN specifically targets JAK2V617F HSCs and if and why it does not have the same effect on CALRm patients.

Our previous clinical study using clonal architecture data combined with a mathematical model indicates that depletion of JAK2V617F HSC by differentiation into progenitors and thus loss of self-renewal may be the critical mechanism for eradication of JAK2V617F disease by IFN. We hope to confirm this hypothesis in a larger number of patients and to understand the basis of the differential effects of JAK2V617F and CALRm mutations on disease-initiating stem cells.

The secondary objectives are to:

* Validate the resistance of CALRm patients to IFN treatment in a larger number of patients. Moreover, high IFN doses, in contrast to JAK2V617F patients, are deleterious to the molecular response for reasons that remain to be understood.
* Investigate the role of associated mutations in IFN-induced molecular responses.

IFN treatments have been shown to promote the appearance of clones (JAK2V617F positive or JAK2V617F negative) with additional mutations, such as Tet2 or DNMT3a, which could be responsible for resistance to IFN treatment . We would like to increase the number of patients and their follow-up to analyze the role of these mutations in treatment success. Moreover, these additional mutations (new or selected by the treatment) could favor the development of more severe pathologies (MF, MDS, AML) than PV or TE and would be important to monitor on the follow-up of IFN-treated patients.

-Explore in vitro the effect of IFN in combination with other molecules on primary patients' cells. Indeed, our basic study already showed the involvement of PML in the mechanism of action of IFN and we found that arsenic greatly potentiates the effect of IFN. We will deeply investigate by which exact mechanisms.

All the data will be collected in patients before IFN treatment or during the IFN treatment and data will be collected by single cell genotyping of colonies and/or by single cell RNA sequencing coupled to genotyping of mutations and/or in vitro assays.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female 18 years of age or older
2. Diagnosis of MPN has been previously established by the referring physician and that physician will have decided to treat with pegylated IFN. Patients will be treated or untreated at the time of inclusion and may be newly diagnosed patients.
3. These patients will be affiliated with or benefit from a social security plan
4. For all these patients an additional 20-40 mL will be collected except for some PV patients who are treated conventionally by phlebotomy. In this case, we will collect blood bags from these patients. The volumes vary between 300 and 450 mL of blood depending on the weight and size of the patients.
5. We will also include in this protocol any patient whose MPN, either PV, TE or MF, will have progressed to acute leukemia (AL) during treatment. These will be patients with AP of MPN (MPN can also progress to acute myeloid leukemia (AML) by acute transformation (AT) of MPN).
6. Patient with signed informed consent

Exclusion Criteria:

1. The non-inclusion criterion concerns the anemia that some MF patients may suffer from. Therefore, patients with anemia (Hb<10g) or transfusion dependency (≥ 1 packed red blood cell per month) at the time of the referral monitoring visit are not included in the research.
2. Persons under court protection, guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The studied population will be all men and women of legal age who were not vulnerable and whose diagnosis of MPN had been previously established by the referring physician. They are therefore voluntary patients of legal age who are not vulnerable and who suffer from PV, ET or MF. The selection of patients is according to the availability of the caregivers for this study but with a preference for this second study towards CALRm patients (rarer) rather than JAK2V617F. Our wish is to integrate a maximum of 50 patients (10/year) knowing that the limitation is the capacity (personnel and finance) of our INSERM laboratory to study this high number of patients.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2028-03-16 (Estimated); Study Completion 2033-03-16 (Estimated)

PRIMARY OUTCOMES:
Clonal architecture of hematopoietic progenitors of patients | During 5 years from day 0 of IFN treatment, 3 to 4 times per year
  Blood samples are processed to separate mature cells (granulocytes) from progenitors (CD34+ marker). Progenitors are isolated and separated by FACS according to their more or less mature CD34+/CD38±/CD90± phenotype and then cultured for 14 days at the single-cell level. The cells resulting from their differentiation in culture are lysed and their DNA is isolated and stored for PCR or NGS analysis in order to define their mutational profile. Once the genotyping of these cells is established, the DNA is destroyed and nothing remains of the initial biological sample.
Single cell RNA sequencing coupled to genotyping | at day 0 of IFN treatment and at two other time point (between 3 and 24 months of treatment)
  Blood samples are processed to separate mature cells (granulocytes) from progenitors (CD34+ marker). Progenitors are isolated and subjected to scRNA-seq using long-read techniques (PromethION). The trajectories of hematopoietic differentiation and RNA sequencing will be analyzed in each cell
Culture of progenitors in vitro | during 5 years from day 0
  Blood samples are processed to separate mature cells (granulocytes) from progenitors (CD34+ marker). Progenitors (CD34+) are then cultured in serum free medium with cytokines or in semisolid medium in the presence of IFN alone or in association.

CONTACTS AND LOCATIONS:
Overall Officials: Florence Pasquier, MD,PhD, Principal Investigator — florence.pasquier@gustaveroussy.fr
Locations (1):
- Inserm U1287, Villejuif, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] James C, Ugo V, Le Couedic JP, Staerk J, Delhommeau F, Lacout C, Garcon L, Raslova H, Berger R, Bennaceur-Griscelli A, Villeval JL, Constantinescu SN, Casadevall N, Vainchenker W. A unique clonal JAK2 mutation leading to constitutive signalling causes polycythaemia vera. Nature. 2005 Apr 28;434(7037):1144-8. doi: 10.1038/nature03546. PMID 15793561
- [Result] Klampfl T, Gisslinger H, Harutyunyan AS, Nivarthi H, Rumi E, Milosevic JD, Them NC, Berg T, Gisslinger B, Pietra D, Chen D, Vladimer GI, Bagienski K, Milanesi C, Casetti IC, Sant'Antonio E, Ferretti V, Elena C, Schischlik F, Cleary C, Six M, Schalling M, Schonegger A, Bock C, Malcovati L, Pascutto C, Superti-Furga G, Cazzola M, Kralovics R. Somatic mutations of calreticulin in myeloproliferative neoplasms. N Engl J Med. 2013 Dec 19;369(25):2379-90. doi: 10.1056/NEJMoa1311347. Epub 2013 Dec 10. PMID 24325356
- [Result] Mascarenhas J, Kosiorek HE, Prchal JT, Rambaldi A, Berenzon D, Yacoub A, Harrison CN, McMullin MF, Vannucchi AM, Ewing J, O'Connell CL, Kiladjian JJ, Mead AJ, Winton EF, Leibowitz DS, De Stefano V, Arcasoy MO, Kessler CM, Catchatourian R, Rondelli D, Silver RT, Bacigalupo A, Nagler A, Kremyanskaya M, Levine MF, Arango Ossa JE, McGovern E, Sandy L, Salama ME, Najfeld V, Tripodi J, Farnoud N, Penson AV, Weinberg RS, Price L, Goldberg JD, Barbui T, Marchioli R, Tognoni G, Rampal RK, Mesa RA, Dueck AC, Hoffman R. A randomized phase 3 trial of interferon-alpha vs hydroxyurea in polycythemia vera and essential thrombocythemia. Blood. 2022 May 12;139(19):2931-2941. doi: 10.1182/blood.2021012743. PMID 35007321
- [Result] Mosca M, Hermange G, Tisserand A, Noble R, Marzac C, Marty C, Le Sueur C, Campario H, Vertenoeil G, El-Khoury M, Catelain C, Rameau P, Gella C, Lenglet J, Casadevall N, Favier R, Solary E, Cassinat B, Kiladjian JJ, Constantinescu SN, Pasquier F, Hochberg ME, Raslova H, Villeval JL, Girodon F, Vainchenker W, Cournede PH, Plo I. Inferring the dynamics of mutated hematopoietic stem and progenitor cells induced by IFNalpha in myeloproliferative neoplasms. Blood. 2021 Dec 2;138(22):2231-2243. doi: 10.1182/blood.2021010986. PMID 34407546
- [Result] Dagher T, Maslah N, Edmond V, Cassinat B, Vainchenker W, Giraudier S, Pasquier F, Verger E, Niwa-Kawakita M, Lallemand-Breitenbach V, Plo I, Kiladjian JJ, Villeval JL, de The H. JAK2V617F myeloproliferative neoplasm eradication by a novel interferon/arsenic therapy involves PML. J Exp Med. 2021 Feb 1;218(2):e20201268. doi: 10.1084/jem.20201268. PMID 33075130
- [Result] Gisslinger H, Klade C, Georgiev P, Krochmalczyk D, Gercheva-Kyuchukova L, Egyed M, Rossiev V, Dulicek P, Illes A, Pylypenko H, Sivcheva L, Mayer J, Yablokova V, Krejcy K, Grohmann-Izay B, Hasselbalch HC, Kralovics R, Kiladjian JJ; PROUD-PV Study Group. Ropeginterferon alfa-2b versus standard therapy for polycythaemia vera (PROUD-PV and CONTINUATION-PV): a randomised, non-inferiority, phase 3 trial and its extension study. Lancet Haematol. 2020 Mar;7(3):e196-e208. doi: 10.1016/S2352-3026(19)30236-4. Epub 2020 Jan 31. PMID 32014125
- [Result] Verger E, Cassinat B, Chauveau A, Dosquet C, Giraudier S, Schlageter MH, Ianotto JC, Yassin MA, Al-Dewik N, Carillo S, Legouffe E, Ugo V, Chomienne C, Kiladjian JJ. Clinical and molecular response to interferon-alpha therapy in essential thrombocythemia patients with CALR mutations. Blood. 2015 Dec 10;126(24):2585-91. doi: 10.1182/blood-2015-07-659060. Epub 2015 Oct 20. PMID 26486786
- [Result] Knudsen TA, Skov V, Stevenson K, Werner L, Duke W, Laurore C, Gibson CJ, Nag A, Thorner AR, Wollison B, Hansen DL, Ellervik C, El Fassi D, de Stricker K, Ocias LF, Brabrand M, Bjerrum OW, Overgaard UM, Frederiksen M, Kristensen TK, Kruse TA, Thomassen M, Mourits-Andersen T, Severinsen MT, Stentoft J, Starklint J, Neuberg DS, Kjaer L, Larsen TS, Hasselbalch HC, Lindsley RC, Mullally A. Genomic profiling of a randomized trial of interferon-alpha vs hydroxyurea in MPN reveals mutation-specific responses. Blood Adv. 2022 Apr 12;6(7):2107-2119. doi: 10.1182/bloodadvances.2021004856. PMID 34507355